CLINICAL TRIAL: NCT04592094
Title: Evaluation of Performances and Safety of the Medical Device Blueback® Physio for Patients With Chronic Low Back Pain
Acronym: ABC-TRACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blueback (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00651-38
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain, Recurrent
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueback® Physio (Experimental): Classic protocole with the use of Blueback® Physio during physiotherapy sessions, , and using the Blueback® Physio in the active mode (patient and physiotherapists see the biofeedback in real time)during the tests required by the protocol of the study.
  Interventions: Device: Blueback® Physio
- Standard Care (No Intervention): Classic protocole without the use of Blueback® Physio during physiotherapy sessions, and using the Blueback® Physio in the blind mode during the tests required by the protocol of the study

INTERVENTIONS:
Device: Blueback® Physio — Blueback® Physio is monitoring the activation level of the transversus abdominis muscle in real time during the exercises
  Arms: Blueback® Physio

SUMMARY:
The main objective of this clinical investigation is to show the superiority of a rehabilitation based on the use of Blueback® Physio compared to a rehabilitation without the use of Blueback® Physio in terms of reducing the time needed for a patient to control the voluntary contraction of the transversus abdominal muscle and to return to autonomy.

DETAILED DESCRIPTION:
The Blueback® Physio is a wireless device for indicating, for a given patient, the relative level of contraction of the transversus abdominal muscle.

Blueback® Physio is a CE marked class I medical device. This medical device allows to measure and visualize in real time the activity of the transversus abdominal muscle, one of the deepest muscle of the abdominal wall. It is placed on the patient, during a rehabilitation session with a mhysiotherapist.

The objective is to optimize the three key phases followed by the healthcare professional: teaching his patient to feel the contraction of the muscle, learning to control this contraction, then learning to master this contraction when the patient is in double task (movements rehabilitation targeting other muscles, cognitive tasks or other tasks of everyday life that strain the spine).

In the ABC-TRACC study, the objective is to compare the time needed for patient to get a good motor control on his transversus abdominal muscle if he is using the Blueback® Physio during his sessons or not.

ELIGIBILITY:
Inclusion Criteria:

* Included in the PRESDO program,
* Suffering from chronic low back pain (= low back pain installed for more than 2 months),
* Beneficiary of a social security,
* For which his consent has been obtained in writing with regard to his participation in the protocol.

Exclusion Criteria:

* Bedridden or using a wheelchair,
* Having a contraindication to performing the muscular exercises provided for in the protocol,
* Having any other condition which, in the opinion of healthcare professionals, could affect its ability to complete the study or could present a significant risk,
* Simultaneously participating in another clinical research protocol or having recently participated in another research for which the exclusion period has not been completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Time needed to master the motor control of the muscle (in number of rehabilitation sessions) | 5 weeks including 5 rehabilitation sessions per week
  The patient is mastering the motor control of the muscle on defined exercises with a quotation calculated using the Blueback Physio.
  The primary outcome measure is a composite between two tests mesauring the ability for the patient to control his mucle activity, and a third test to measure his autonomy on this control (does the patient has enough awarness of his own ability to control the muscle).
  The three tests are underwent using the Blueback Physio in order th get the quotations used for the calculations.

SECONDARY OUTCOMES:
Well-being for daily life based on a questionnaire | 5 weeks
  This secondary outcome will be assessed by using the NHP questionnaire. Each section of the questionnaire is rated between 0 and 100. A higher rate shows a lower well-being for the patient.
Well-being for daily life based on a muscular test | 5 weeks
  This secondary outcome will be assessed by using a muscular test (ito-shirado and sorensen). The tests consist in calculating the time during which the patient can maintain the requested posture. THe outcome is evaluated by calculating the ratio between the two tests. The closer to one (value 1) the better.
Pain feeling | 5 weeks
  This secondary criteria will be assessed using the NHP questionnaire. Each section of the questionnaire is rated between 0 and 100. A higher rate shows a lower well-being for the patient.
Medical Device Safety | 5 weeks
  The MD safety will be assessed by analysing the Undesirable side-effects and the Defects reported during the investigation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin MARGO, MD, Principal Investigator — Centre Médical et Pédagogique de Beaulieu
Locations (1):
- Clinique FSEF Rennes BEAULIEU, Rennes, France

IPD SHARING:
Plan to Share IPD: No